CLINICAL TRIAL: NCT02955212
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study With Upadacitinib (ABT-494) in Subjects From China and Selected Countries With Moderately to Severely Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Conventional Synthetic Disease-Modifying Anti-Rheumatic Drugs (csDMARDs)
Brief Title: A Study With Upadacitinib (ABT-494) in Subjects From China and Selected Countries With Moderately to Severely Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Conventional Synthetic Disease-Modifying Anti-Rheumatic Drugs (csDMARDs)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-557
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-08

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis; Conventional Synthetic Disease-Modifying Anti-Rheumatic Drugs (csDMARDs); ABT-494
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo / Upadacitinib 15 mg (Placebo Comparator): Participants randomized to receive placebo once daily for 12 weeks in Period 1 followed by upadacitinib 15 mg once daily for up to 52 weeks in Period 2.
  Interventions: Drug: Upadacitinib; Drug: Placebo
- Upadacitinib 15 mg (Experimental): Participants randomized to receive upadacitinib 15 mg once daily for 12 weeks in Period 1 and up to an additional 52 weeks in Period 2.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Tablets for oral administration
  Other Names: ABT-494; RINVOQ™
Drug: Placebo — Tablets for oral administration
  Arms: Placebo / Upadacitinib 15 mg

SUMMARY:
The study objectives of Period 1 of this study were to compare the efficacy, safety, and tolerability of upadacitinib versus placebo for the treatment of signs and symptoms of subjects from China and selected countries including Brazil and South Korea with moderately to severely active rheumatoid arthritis (RA) who are on a stable dose of csDMARDs and have an inadequate response to csDMARDs.

The study objective of Period 2 is to evaluate the long-term safety, tolerability, and efficacy of upadacitinib in subjects with RA who have completed Period 1.

DETAILED DESCRIPTION:
This is a Phase 3 multicenter study that includes two periods. Period 1 is a 12-week, randomized, double-blind, parallel-group, placebo-controlled period designed to compare the safety and efficacy of upadacitinib versus placebo for the treatment of signs and symptoms of participants with moderately to severely active RA who are on a stable dose of csDMARDs and have an inadequate response to csDMARDs. Period 2 is an open label 52 week extension period to evaluate the long-term safety, tolerability, and efficacy of upadacitinib in participants with RA who have completed Period 1.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA for ≥ 3 months who also fulfill the 2010 American College of Rheumatology (ACR)/ European League Against Rheumatism (EULAR) classification criteria for RA.
* Participants have been receiving csDMARD therapy ≥ 3 months and on a stable dose for ≥ 4 weeks prior to the first dose of study drug.

  1. Participants must have failed (lack of efficacy) at least one of the following: methotrexate (MTX), sulfasalazine, or leflunomide.
  2. The following csDMARDs are allowed: oral or parenteral MTX, sulfasalazine, hydroxychloroquine, chloroquine, and leflunomide.
  3. A combination of up to two background csDMARDs is allowed except the combination of MTX and leflunomide.
* Participant meets both of the following disease activity criteria:

  1. ≥ 6 swollen joints (based on 66 joint counts) and ≥ 6 tender joints (based on 68 joint counts) at Screening and Baseline Visits; and
  2. High-sensitivity C-Reactive Protein (hsCRP) ≥ 3 mg/L at Screening
* Participants with prior exposure to at most one biological disease-modifying anti-rheumatic drugs (bDMARD) may be enrolled (up to 20% of total number of subjects). Specifically, prior to enrollment:

  1. Participants with limited exposure to bDMARD (< 3 months) OR
  2. Participants who are responding to a bDMARD therapy but had to discontinue due to intolerability (regardless of treatment duration).
* Participants must have discontinued bDMARD therapy prior to the first dose of study drug.

Exclusion Criteria:

* Prior exposure to any Janus kinase (JAK) inhibitor (including but not limited to tofacitinib, baricitinib, and filgotinib).
* Participants who are considered inadequate responders (lack of efficacy) to bDMARD therapy as defined by the Investigator.
* History of any arthritis with onset prior to age 17 years or current diagnosis of inflammatory joint disease other than RA (including but not limited to gout, systemic lupus erythematosus, psoriatic arthritis, axial spondyloarthritis including ankylosing spondylitis and non-radiographic axial spondyloarthritis, reactive arthritis, overlap connective tissue diseases, scleroderma, polymyositis, dermatomyositis, fibromyalgia [currently with active symptoms]. Current diagnosis of secondary Sjogren's Syndrome is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2020-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (43):
- Brazil (5):
  - Ceti - Centro de Estudos Em Terapias Inovadoras Ltda /Id# 152964, Curitiba, Paraná
  - Parana Medical Research Center /ID# 153507, Maringá, Paraná
  - LMK Sevicos Medicos S/S /ID# 152963, Porto Alegre, Rio Grande do Sul
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto /ID# 152961, São José do Rio Preto, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica e Serviços Médicos Ltda /ID# 152966, São Paulo, São Paulo
- China (23):
  - 1st Aff Hosp of Bengbu Med Col /ID# 162161, Bengbu, Anhui
  - Anhui Provincial Hospital /ID# 161117, Hefei, Anhui
  - Zhongshan Hosp. of Fudan Uni. /ID# 161108, Shanghai, Anhui
  - The 1st Aff Hosp Xiamen Univ /ID# 162154, Xiamen, Fujian
  - Zhuzhou Central Hospital /ID# 162153, Zhuzhou, Hunan
  - The First Affiliated Hospital /ID# 163747, Baotou, Inner Mongolia
  - The First People's Hospital /ID# 168462, Changzhou, Jiangsu
  - The First People's Hospital of Jiujiang /ID# 168461, Jiujiang, Jiangxi
  - The First Hosp of Jilin Univ /ID# 161116, Changchun, Jilin
  - Jining No.1 People's Hospital /ID# 162158, Jining, Shandong
  - Shanghai Changhai Hospital /ID# 161123, Shanghai, Shanghai Municipality
  - West China Hospital /ID# 161119, Chengdu, Sichuan
  - Xuanwu Hosp Capital Med Univ /ID# 161118, Beijing
  - Peking Union Med College Hosp /ID# 161107, Beijing
  - The Second Xiangya Hospital of Central South University /ID# 162152, Changsha
  - First Affiliated Hospital of Kunming Medical University /ID# 164637, Kunming
  - Jiangsu Province Hospital /ID# 161122, Nanjing
  - Pingxiang People's Hospital /ID# 162151, Pingxiang
  - 1st Aff Hosp of Shantou Univ /ID# 162165, Shantou Guangdong
  - The Second Hospital of Shanxi /ID# 162164, Taiyuan
  - Tianjin Med Univ General Hosp /ID# 162155, Tianjin
  - People's Hospital of Xinjiang /ID# 162157, Ürümqi
  - First Affiliated Hospital of Xi'an Jiaotong University /ID# 162150, Xi'an
- South Korea (15):
  - SoonChunHyang University CheonAn Hospital /ID# 209078, Cheonan-si, Chungcheongnam-do
  - Kyungpook National Univ Hosp /ID# 166919, Daegu, Daegu Gwang Yeogsi
  - Chungnam National University Hospital /ID# 167727, Junggu, Daejeon Gwang Yeogsi
  - St. Vincent's Hospital /ID# 166918, Suwon, Gyeonggido
  - Ajou University Hospital /ID# 163912, Suwon, Gyeonggido
  - Inha University Hospital /ID# 163910, Junggu, Incheon Gwang Yeogsi
  - Chonnam National University Hospital /ID# 167726, Gwangju, Jeonranamdo
  - Kyung Hee University Medical Center /ID# 163908, Dongdaemun-gu, Seoul Teugbyeolsi
  - SMG-SNU Boramae Medical Center /ID# 163911, Dongjak-gu, Seoul Teugbyeolsi
  - Yonsei University Health System, Severance Hospital /ID# 168421, Seodaemun-gu, Seoul Teugbyeolsi
  - Hanyang University Seoul Hospi /ID# 163913, Seongdong-gu, Seoul Teugbyeolsi
  - Konkuk University Medical Ctr /ID# 206148, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Yeouido St. Mary's Hospital /ID# 204224, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 163909, Seoul
  - Chung-Ang University Hostipal /ID# 209076, Seoul

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 37 sites in Brazil, China, and South Korea.
  The study consisted of a 12-week placebo-controlled, double-blind period (Period 1), and an open-label 52-week extension period (Period 2).
Pre-assignment Details: Participants who met eligibility criteria were randomized in a 1:1 ratio to one of two treatment groups. Randomization was stratified by country and the Chinese population was expected to comprise up to 80% of the total study population.
Groups:
- Upadacitinib 15 mg / Upadacitinib 15 mg: Participants randomized to receive upadacitinib 15 mg once daily for 12 weeks in Period 1 followed by upadacitinib 15 mg once daily for up to 52 weeks in Period 2.
Period: Period 1: Double-blind Treatment Period
Arm/Group | Placebo / Upadacitinib 15 mg | Upadacitinib 15 mg / Upadacitinib 15 mg
Started | 169 | 169
Completed (Completed Period 1 (Week 12) study drug) | 153 | 157
Not Completed | 16 | 12
Not completed — Adverse Event | 4 | 7
Not completed — Withdrawal by Subject | 8 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 3 | 2
Period: Period 2: Open-label Extension
Arm/Group | Placebo / Upadacitinib 15 mg | Upadacitinib 15 mg / Upadacitinib 15 mg
Started | 153 | 157
Completed | 136 | 139
Not Completed | 17 | 18
Not completed — Adverse Event | 11 | 7
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lack of Efficacy | 3 | 2
Not completed — COVID-19 Logistical Restrictions | 0 | 1
Not completed — Other | 2 | 4

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo: Participants randomized to receive placebo once daily for 12 weeks in Period 1.
- Upadacitinib 15 mg: Participants randomized to receive upadacitinib 15 mg once daily for 12 weeks in Period 1.
- Total: Total of all reporting groups
Arm/Group | Placebo | Upadacitinib 15 mg | Total
Number analyzed (Participants) | 169 | 169 | 338
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (11.39) | 51.7 (10.63) | 51.7 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 135 | 274
  Male | 30 | 34 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 24 | 45
  Not Hispanic or Latino | 148 | 145 | 293
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19 | 19 | 38
  Black or African American | 3 | 3 | 6
  American Indian/Alaska Native | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Asian | 142 | 141 | 283
  Multiple | 5 | 6 | 11
Enrollment by Country [Count of Participants; unit: Participants]
  China | 114 | 114 | 228
  South Korea | 29 | 29 | 58
  Brazil | 26 | 26 | 52
Duration Since Rheumatoid Arthritis (RA) Diagnosis [Mean (Standard Deviation); unit: years] | 7.5 (7.55) | 7.2 (7.16) | 7.3 (7.35)
Tender Joint Count [Mean (Standard Deviation); unit: joints] — A total of 68 joints were assessed for the presence or absence of tenderness.
  joints | 23.0 (14.45) | 21.5 (14.84) | 22.3 (14.64)
Swollen Joint Count [Mean (Standard Deviation); unit: joints] — A total of 66 joints were assessed for the presence or absence of swelling.
  joints | 11.9 (6.00) | 11.9 (6.89) | 11.9 (6.45)
Patient's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: units on a scale] — The participant was asked to rate their current RA disease activity over the past 24 hours on a visual analog scale (VAS) ranging from 0 to 100, where 0 indicates very low disease activity and 100 indicates very high disease activity. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 166 | 166 | 332
    (all) | 63.9 (22.32) | 64.4 (20.52) | 64.1 (21.41)
Physician's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: units on a scale] — The physician rated the participant's current global RA disease activity (independently from the participant's assessment) on a VAS scale from 0 to 100, where 0 indicates very low disease activity and 100 indicates very high disease activity. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 166 | 163 | 329
    (all) | 67.0 (13.83) | 66.7 (17.51) | 66.9 (15.74)
Patient's Assessment of Pain [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to indicate the severity of their arthritis pain within the previous week on a visual analog scale from 0 to 100. A score of 0 indicates "no pain" and a score of 100 indicates "worst possible pain." Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 166 | 165 | 331
    (all) | 63.8 (20.62) | 66.8 (20.59) | 65.3 (20.63)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 166 | 166 | 332
    (all) | 1.4 (0.65) | 1.3 (0.66) | 1.3 (0.65)
High-sensitivity C-reactive Protein (CRP) [Mean (Standard Deviation); unit: mg/L] | 20.2 (25.15) | 20.0 (21.46) | 20.1 (23.34)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom ACR data were missing at Week 12 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 169 | 169
percentage of participants | 31.4 [24.4 to 38.4] | 71.6 [64.8 to 78.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for the stratification factor of country; Response Rate Difference = 40.2, 95% CI 2-sided [30.5 to 50.0] — Response Rate Difference = Upadacitinib - Placebo

2. Secondary Outcome: Change From Baseline in Disease Activity Score Based on CRP (DAS28 [CRP]) at Week 12
Description: The DAS28 (CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to 10, where higher scores indicate more disease activity. A negative change from Baseline in DAS28 (CRP) indicates improvement in disease activity.
Time Frame: Baseline and Week 12
Population: Full analysis set; multiple imputation was used for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 169 | 169
units on a scale | -0.95 [-1.16 to -0.74] | -2.56 [-2.76 to -2.36]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model including treatment as the fixed factor, and Baseline value and the stratification factor country as the covariates; Least Squares (LS) Mean Difference = -1.61, 95% CI 2-sided [-1.86 to -1.36] — LS Mean Difference = Upadacitinib - Placebo

3. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability.
  A negative change from Baseline in the overall score indicates improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set; multiple imputation was used for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 169 | 169
units on a scale | -0.18 [-0.28 to -0.09] | -0.62 [-0.71 to -0.54]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.44, 95% CI 2-sided [-0.55 to -0.33] — LS Mean Difference = Upadacitinib - Placebo

4. Secondary Outcome: Change From Baseline in Short-Form 36 (SF-36) Physical Component Score (PCS) at Week 12
Description: The Short Form 36-Item Health Survey (SF-36) Version 2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical component score is a weighted combination of the 8 subscales with positive weighting for physical functioning, role-physical, bodily pain, and general health. The PCS was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from baseline score indicates an improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available data; a mixed effect model repeat measurement (MMRM) analysis with data from observed cases to Week 12 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 149 | 143
units on a scale | 3.36 [2.25 to 4.48] | 8.93 [7.80 to 10.07]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; MMRM model with treatment, visit, treatment-by-visit interaction and stratification factor of country as fixed effects and Baseline value as covariate; LS Mean Difference = 5.57, 95% CI 2-sided [4.13 to 7.01] — LS Mean Difference = Upadacitinib - Placebo

5. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on DAS28 (CRP) at Week 12
Description: Low disease activity based on DAS28 (CRP) is defined a DAS28 (CRP) score of ≤ 3.2.
  The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to 10, where higher scores indicate more disease activity. A DAS28 score less than or equal to 3.2 indicates low disease activity.
Time Frame: Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom DAS28 data were missing at Week 12 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 169 | 169
percentage of participants | 13.6 [8.4 to 18.8] | 46.2 [38.6 to 53.7]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for the stratification factor country; Response Rate Difference = 32.5, 95% CI 2-sided [23.4 to 41.7] — Response Rate Difference = Upadacitinib - Placebo

6. Secondary Outcome: Percentage of Participants Achieving Clinical Remission Based on DAS28 (CRP) at Week 12
Description: Clinical remission (CR) based on DAS28 (CRP) is defined as achieving a DAS28 (CRP) score of less than 2.6.
  DAS28 (CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to 10, where higher scores indicate more disease activity.
Time Frame: Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom DAS28 (CRP) data were missing at Week 12 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 169 | 169
percentage of participants | 5.3 [1.9 to 8.7] | 29.6 [22.7 to 36.5]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for the stratification factor of country; Response Rate Difference = 24.3, 24.3% CI 2-sided [16.6 to 31.9] — Response Rate Difference = Upadacitinib - Placebo

7. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity Based on Clinical Disease Activity Index (CDAI) at Week 12
Description: Low disease activity based on CDAI is defined as a CDAI score ≤ 10. CDAI is a composite index for assessing disease activity based on the summation of the total tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 76 with higher scores indicating higher disease activity.
Time Frame: Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom CDAI data were missing at Week 12 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 169 | 169
percentage of participants | 11.2 [6.5 to 16.0] | 35.5 [28.3 to 42.7]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for the stratification factor of country; Response Rate Difference = 24.3, 95% CI 2-sided [15.6 to 32.9] — Response Rate Difference = Upadacitinib - Placebo

8. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 169 | 169
percentage of participants | 8.3 [4.1 to 12.4] | 40.8 [33.4 to 48.2]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for the stratification factor of country; Response Rate Difference = 32.5, 95% CI 2-sided [24.0 to 41.0] — Response Rate Difference = Upadacitinib - Placebo

9. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR70 response criteria:
  1. ≥ 70% improvement in 68-tender joint count;
  2. ≥ 70% improvement in 66-swollen joint count; and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 169 | 169
percentage of participants | 3.6 [0.8 to 6.3] | 21.3 [15.1 to 27.5]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for the stratification factor of country; Response Rate Difference = 17.8, 95% CI 2-sided [11.0 to 24.5] — Response Rate Difference = Upadacitinib - Placebo

10. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 1
Description: as for outcome 1
Time Frame: Baseline and Week 1
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 1 or for whom ACR data were missing at Week 1 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg
Number analyzed (Participants) | 169 | 169
percentage of participants | 5.9 [2.4 to 9.5] | 25.4 [18.9 to 32.0]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for the stratification factor of country; Response Rate Difference = 19.5, 95% CI 2-sided [12.1 to 27.0] — Response Rate Difference = Upadacitinib - Placebo

ADVERSE EVENTS:
Time Frame: Period 1: From the first dose of study drug up to Week 12 or up to 30 days after last dose for participants who discontinued study drug prior to Week 12. Period 2: From Week 12 to 30 days after last dose; up to 56 weeks.
Groups:
- Period 1: Placebo: Participants received placebo once daily for 12 weeks in Period 1.
- Period 1: Upadacitinib 15 mg: Participants received upadacitinib 15 mg once daily for 12 weeks in Period 1.
- Period 1+2: Upadacitinib 15 mg: Participants originally assigned to placebo received upadacitinib 15 mg from Week 12 to Week 64. Participants originally assigned to upadacitinib received upadacitinib 15 mg from Week 0 to Week 64.
Arm/Group | Period 1: Placebo | Period 1: Upadacitinib 15 mg | Period 1+2: Upadacitinib 15 mg
All-Cause Mortality (participants affected / at risk) | 0/169 | 0/169 | 0/322
Serious Adverse Events (participants affected / at risk) | 5/169 | 12/169 | 55/322
Other Adverse Events (participants affected / at risk) | 13/169 | 25/169 | 198/322
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Placebo (N=169) | Period 1: Upadacitinib 15 mg (N=169) | Period 1+2: Upadacitinib 15 mg (N=322)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1) | 4 (4)
PNEUMONIA (Infections and infestations) | 1 (1) | 3 (3) | 8 (8)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (3)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
SENILE OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SPINAL LIGAMENT OSSIFICATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
URETEROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
DUODENAL ULCER PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
FALLOPIAN TUBE ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
FEBRILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA CRYPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
SINUSITIS FUNGAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
ACOUSTIC NEUROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
KAPOSI'S SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA OF THE CERVIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
POST HERPETIC NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
ABORTION INDUCED (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Placebo (N=169) | Period 1: Upadacitinib 15 mg (N=169) | Period 1+2: Upadacitinib 15 mg (N=322)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 (13) | 16 (16) | 65 (95)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 9 (13) | 30 (43)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 26 (30)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 26 (37)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 20 (27)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 (0) | 0 (0) | 27 (34)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 23 (24)
LATENT TUBERCULOSIS (Infections and infestations) | 0 (0) | 0 (0) | 18 (18)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 24 (29)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 19 (21)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 24 (33)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 0 (0) | 29 (37)
WEIGHT INCREASED (Investigations) | 0 (0) | 0 (0) | 23 (31)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT02955212/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT02955212/SAP_001.pdf